CLINICAL TRIAL: NCT03480191
Title: Adjunction of Daptomycin for the Treatment of Pneumococcal Meningitis: AddaMAP Study
Brief Title: Adjunction of Daptomycin for the Treatment of Pneumococcal Meningitis
Acronym: AddaMAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAVANET-PHRC-2016
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Meningitis
MeSH Terms: conditions — Meningitis, Pneumococcal | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — Daptomycin will be given by intravenous infusion and administered over a 30 minutes infusion, daily, for 8 days and at the dosis of 10mg/kg/day.

SUMMARY:
Pneumococcal meningitis is an infection of the membrane that covers the brain. It is a serious infection which is currently treated with a combination of corticosteroids (dexamethasone) and 3rd generation cephalosporins. Nevertheless, complications associated with meningitis are relatively frequent and severe. Recent animal studies have shown that another antibiotic, daptomycin, can reduce the mortality and long-term effects of pneumococcal meningitis. Daptomycin is widely used worldwide in humans for other diseases, with few side effects.

This study aims to evaluate the effect of daptomycin on the proliferation of the bacterial infection, and therefore on inflammation. Daptomycin will be added to the currently recommended treatment with the same dosage used for other diseases.

Roughly 130 patients with suspected pneumococcal meningitis admitted to the emergency departments of hospitals throughout France will be asked to participate in this study.

The participation period will last approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged over 18 years
* With Suspected pneumococcal meningitis :

  * clinical presentation evocative of pneumococcal meningitis : acute onset of ,meningeal signs, history of cranial trauma or fistula, knowledge of alteration of humoral immunity,, asplenia, alcoholism with/or
  * clearly purulent CSF with/ or,
  * presence of diplococcus on the Gram stain of CSF or positive pneumococcal antigen in the CSF, or polymorphonuclear cells in CSF > 100
* Written consent or inclusion in an emergency
* Affiliation to a social security system

Exclusion Criteria:

* Contraindication to cephalosporin
* Immediate and severe hypersensitivity to β-lactam antimicrobial
* Contraindication to dexamethasone
* Contraindication to daptomycin
* Previous exposition to daptomycin (within one year)
* Women who are able to procreate without effective contraception and pregnant or breastfeeding women
* Patients under ward of court
* Refusal at any time after acceptation of the study from the patient or her/his legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Disability-free survival, assessed with the modified Rankin Scale (mRS) | At Day 30

SECONDARY OUTCOMES:
Overall mortality | At Day 30 and Day 90
Disability level assessed with the mRS in surviving patients | At Day 30 and Day 90
Disability level assessed with the Glascow Coma Scale and the Glasgow Outcome Scale in the overall efficacy population | At Day 30 and Day 90
Disability level assessed with mini-mental score in surviving patients | At Day 30 and Day 90
Hearing loss assessed with the Hearing Handicap Inventory test | At Day 30 and Day 90
Hearing loss assessed with audiometry | At Day 30
Hearing loss assessed with the Hearing-it test | At Day 30
Quality of life assessed with the 12-Item Short Form Health Survey (SF-12) | At Day 30 and Day 90
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Quality of life assessed with WHO QOL BREF | At Day 30 and Day 90
Number of days without hospitalisation (including ICU) | At Day 30 and Day 90
Number of days without antimicrobial therapy | At Day 30
Frequency and type of side effects related to daptomycine | Within 30 days after daptomycin start

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
the study team is available to collaborate with other research teams on reasonable request to access study data

REFERENCES:
- [Derived] Chavanet P, Fournel I, Bourredjem A, Piroth L, Blot M, Sixt T, Binquet C. Addition of daptomycin for the treatment of pneumococcal meningitis: protocol for the AddaMAP study. BMJ Open. 2023 Jul 25;13(7):e073032. doi: 10.1136/bmjopen-2023-073032. PMID 37491088
- [Derived] Wall EC, Chan JM, Gil E, Heyderman RS. Acute bacterial meningitis. Curr Opin Neurol. 2021 Jun 1;34(3):386-395. doi: 10.1097/WCO.0000000000000934. PMID 33767093